CLINICAL TRIAL: NCT04057807
Title: PBR28 Brain Positron Emission Tomography Imaging With Lipopolysaccharide (LPS) Challenge for the Study of Microglia Function in Alzheimer's Disease
Brief Title: Peripheral Benzodiazepine Receptors (PBR28) Brain PET Imaging With Lipopolysaccharide Challenge for the Study of Microglia Function in Alzheimer's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1611018611; 1K23AG057794-01 (NIH)
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients receiving endotoxin (Experimental): The 20 enrolled subjects will have LPS (0.4 ng/kg) administered intravenously
  Interventions: Drug: LPS

INTERVENTIONS:
Drug: LPS — LPS (0.4 ng/kg)

SUMMARY:
To examine the differences in the capacity to activate microglia in patients with Alzheimer's Disease (AD) compared to age-comparable cognitively normal subjects and younger healthy controls.

DETAILED DESCRIPTION:
The primary outcome is Microglia Activation Reserve Index (MARI) (calculated in the parietal region of interest (ROIs)) in AD patients compared to elderly controls. The researchers will recruit up to 20 participants. The investigators will use 7 AD and 7 comparably aged cognitively normal successfully scanned subjects to calculate the microglial activation reserve index. The expectations are significant differences between the two groups suggesting altered reactivity of the microglia in AD. The result would be an exciting one suggesting at least one mechanism by which some patients with significant amyloid load have progressive dementia while comparable others are either cognitively normal or have stable Mild Cognitive Impairment (MCI). It will also suggest avenues for intervention in amyloid positive MCIs to prevent progression to Alzheimer's dementia. The exploratory analysis will include:

1. Effects of aging on MARI: The researchers will evaluate the effects of aging on MARI. Comparisons will be made for MARI between cognitively normal elderly and the 8 healthy individuals to whom the investigators applied this protocol in an earlier study. The reactivity of microglia is reported to change with age and so the investigators expect MARI to change in the cognitively normal elderly. However, the expectation is that the differences between the young and elderly cognitively normal subjects to be small relative to the comparison of AD and elderly normal controls.
2. Effects of amyloid on MARI: The researchers will look at the relationship of regional and global amyloid load to MARI. The presence of a relationship suggests that one of the reasons for altered microglial reactivity might be interactions of microglia with pathologic amyloid.
3. Effects of MARI on cognition: The researchers will explore whether MARI would correlate with the measure of disease stage, with higher MARIs associated with worse neuropsychological score and more severe disease. The researchers will look for correlations between MARI and the individual neuropsychological scores. This would determine if disease severity is correlated with microglial activation reserve.

ELIGIBILITY:
Inclusion Criteria:

* Mild AD Subjects:
* National Institute on Aging (NIA)-Alzheimer's Association core clinical criteria for probable AD
* Age between 55 and 90 (inclusive)
* Score on the Montreal Cognitive Assessment (MOCA) greater than or equal to 17
* Presence of a responsible caregiver who will accompany AD subjects to all procedures.
* Biomarker evidence of Alzheimer's disease via an amyloid PET scan or cerebrospinal fluid (CSF) amyloid Beta measurement.
* The patient should have the capacity to consent.
* Clinical Dementia Rating (CDR) global score greater than 0.
* Cognitively normal elderly Subjects:
* Absence of National Institute on Aging-Alzheimer's Association core clinical criteria for probable AD
* Objective memory scores within the normal range for age (do not meet MCI Subjects criterion 2)
* Age between 55 and 90 (inclusive)
* Clinical Dementia Rating (CDR) global score of 0.0

Exclusion Criteria:

* Any significant neurologic disease (other than probable AD in the AD Subjects group), such as stroke, Parkinson's disease, brain tumor, seizure disorder, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits.
* Any significant systemic disease including hepatic failure, heart failure, renal failure, chronic obstructive pulmonary disease (COPD), active infection and autoimmune disease.
* Screening/baseline MRI scan with evidence of infection, infarction, or other focal lesions. Subjects with multiple lacunes or lacunes in a critical memory structure are excluded.
* Any significant systemic illness or unstable medical condition, including uncontrolled or insulin- dependent diabetes mellitus, uncorrected hypothyroidism or hyperthyroidism, or systemic cancer.
* Current or regular use of over-the-counter medication that may affect the immune system (e.g., ibuprofen), including corticosteroids or immunosuppressant drugs; no use in 3 weeks prior to the PET scan
* Investigational agents are prohibited 4 weeks prior to entry and for the duration of the study.
* Previous treatment with an investigational small molecule with anti-amyloid properties or passive immunization against amyloid within 1 year of study entry.
* Previous treatment with an active immunization against amyloid.
* History of schizophrenia or other major psychiatric disorder (DSM IV criteria).
* History of alcohol or substance abuse or dependence (DSM IV criteria) within the past 2 years.
* Clinically significant abnormalities on screening laboratory tests (B12, Thyroid function tests, hematology, chemistry, urinalysis, ECG).
* Pregnancy, as determined by screening pregnancy tests for pre-menopausal females
* Impairment of visual or auditory acuity sufficient to interfere with study procedures.
* Education level < 6 years.
* Evidence of current depression as defined by a score of ≥ 5 on the Geriatric Depression Scale.
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body. The presence of claustrophobia, precluding MRI.
* Current or recent participation in any procedures involving radioactive agents such that the total radiation dose exposure to the subject in any given year would exceed the limits of annual and total dose commitment set forth in the US Code of Federal Regulations (CFR) Title 21 Section 361.1.
* Vaccination in the last month.
* Drink more than 5 alcoholic drinks per week or any heavy drinking days in the last 30 days.
* BMI > 35 or < 19
* Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or Intrauterine Device (IUD)
* Individuals who are classified as "low binders" for the rs6971 polymorphism (<10% of the population)
* Patients on antiplatelet and anticoagulant medications will be excluded.
* Any patient without the capacity to consent will be excluded.
* Unstable hypertension. If blood pressure is greater than 160/100, the investigators will contact the subject's primary care physician to manage their blood pressure. If their blood pressure is not reduced to be consistently below 160/100 by the scanning day the subject will be excluded from the protocol.
* Patients with contraindications for lumbar puncture procedure can be still involved and will be excluded from the optional portion of the study with the lumbar puncture. These include existing intracranial space-occupying lesion with mass effect, posterior fossa mass, risk of cerebral herniation by increased CSF pressure or Arnold chiari malformation, as well as anticoagulant medication, coagulopathies and uncorrected bleeding diathesis, congenital spine abnormalities, and local skin infection at the puncture site.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Mecca, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- Alzheimer's Disease Research Unit, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Receiving Endotoxin: The enrolled subjects will have LPS (0.4 ng/kg) administered intravenously
  LPS: LPS (0.4 ng/kg)
Period: Overall Study
Arm/Group | Patients Receiving Endotoxin
Started | 12
1 Week Follow up | 11 (1 participant did not receive one week follow up (missed visit), resumed at 6 month follow up)
6 Month Follow up | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Receiving Endotoxin: The enrolled subjects, both with AD and cognitively normal, will have LPS (0.4 ng/kg) administered intravenously
  LPS: LPS (0.4 ng/kg)
Arm/Group | Patients Receiving Endotoxin
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline measures were collected by cognitive status.
  years
    Alzheimer's Disease: number analyzed (Participants) | 6
    Alzheimer's Disease | 75.3 (2.3)
    Cognitively Normal: number analyzed (Participants) | 6
    Cognitively Normal | 67.2 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline measures were collected by cognitive status.
  Participants
    Alzheimer's Disease: number analyzed (Participants) | 6
    Alzheimer's Disease: Female | 1
    Alzheimer's Disease: Male | 5
    Cognitively Normal: number analyzed (Participants) | 6
    Cognitively Normal: Female | 3
    Cognitively Normal: Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline measures were collected by cognitive status.
  Participants
    Alzheimer's Disease: number analyzed (Participants) | 6
    Alzheimer's Disease: White | 6
    Alzheimer's Disease: Black | 0
    Cognitively Normal: number analyzed (Participants) | 6
    Cognitively Normal: White | 5
    Cognitively Normal: Black | 1
Region of Enrollment [Number; unit: participants]
  United States | 12
Global Clinical Dementia Rating Global Score (CDR) [Mean (Standard Deviation); unit: score on a scale] — CDR rates 6 domains of functioning: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a 5-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). The global score is obtained by summing each of the domain box scores, with scores ranging from 0 to 18. Higher scores indicate more severe dementia. Population: Baseline measures were collected by cognitive status.
  score on a scale
    Alzheimer's Disease: number analyzed (Participants) | 6
    Alzheimer's Disease | 0.75 (0.27)
    Cognitively Normal: number analyzed (Participants) | 6
    Cognitively Normal | 0 (0)
Montreal Cognitive Assessment (MOCA) [Mean (Standard Deviation); unit: score on a scale] — MOCA is a brief, useful and validated cognitive screening instrument to differentiate mild cognitive impairment (MCI) or dementia from normal. Range of total score 0-30 where higher scores represent better cognitive performance. Population: Baseline measures were collected by cognitive status.
  score on a scale
    Alzheimer's Disease: number analyzed (Participants) | 6
    Alzheimer's Disease | 21.5 (3.8)
    Cognitively Normal: number analyzed (Participants) | 6
    Cognitively Normal | 26.7 (2.4)
Number of participants with one of two rs6971 polymorphism [Count of Participants; unit: Participants] — To determine which rs6971 polymorphism is present in the two cognitive states. Population: Baseline measures were collected by cognitive status.
  Participants
    Alzheimer's Disease: number analyzed (Participants) | 6
    Alzheimer's Disease: mixed affinity binder (MAB) | 0
    Alzheimer's Disease: high affinity binder (HAB) | 6
    Cognitively Normal: number analyzed (Participants) | 6
    Cognitively Normal: mixed affinity binder (MAB) | 3
    Cognitively Normal: high affinity binder (HAB) | 3

OUTCOME MEASURES:

1. Primary Outcome: Microglial Activation Reserve Index (MARI)
Description: Participants will undergo [11C]PBR PET scanning both before and then after LPS injection. Parametric images of volume of distribution (VT)were generated for each using multilinear analysis (MA1) and MARI was calculated in the parietal cortex using the equation [(VT post LPS - VT pre LPS)/VT post LPS] x 100%. Higher values of MARI are thought to represent higher levels of microglial activation. There are no clinically relevant thresholds for this measure.
Time Frame: 180 minutes post intervention
Population: One participant from the cognitively normal group was excluded from this analysis since blood input function data for the baseline scan was inadequate for pharmacokinetic modeling.
Measure: Mean (Standard Deviation); unit: percentage of MARI
Arm/Group | Patients Receiving Endotoxin
Number analyzed (Participants) | 11
percentage of MARI
  Alzheimer's Disease: number analyzed (Participants) | 6
  Alzheimer's Disease | 17.7 (0.1)
  Cognitively Normal: number analyzed (Participants) | 5
  Cognitively Normal | 30.1 (0.1)
Statistical Analysis 1: Comparison: Patients Receiving Endotoxin; Test type: Superiority; p = 0.14, unpaired t-tests (continuous variables)

2. Secondary Outcome: Effects of MARI on Cognition
Description: The Pearson's correlation between MARI and performance on the Montreal Cognitive Assessment (MOCA) will be calculated. The MOCA is a global assessment of cognitive function ranging from 0 to 30 where higher scores represent better cognitive performance.
Time Frame: 180 minutes post intervention
Population: Data are from correlation between parietal cortex MARI and MOCA scores for participants with AD
Measure: Number; unit: Pearson r
Arm/Group | Patients Receiving Endotoxin
Number analyzed (Participants) | 6
Pearson r | -0.12
Statistical Analysis 1: Comparison: Patients Receiving Endotoxin; Test type: Superiority; p = 0.82, univariate linear regression analysis; two-tailed P value was obtained from a univariate linear regression analysis

ADVERSE EVENTS:
Time Frame: 180 minutes post intervention
Arm/Group | Patients Receiving Endotoxin
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04057807/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04057807/ICF_001.pdf